CLINICAL TRIAL: NCT00338988
Title: A Phase II Study of Oxaliplatin and Capecitabine in Patients With Unresectable Cholangiocarcinoma, Including Carcinoma of the Gallbladder and Biliary Tract
Brief Title: Oxaliplatin and Capecitabine in Patients With Unresectable Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0340
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cancer of the Gallbladder; Cancer of the Biliary Tract
Keywords: Gastrointestinal; Capecitabine; Oxaliplatin; Carcinoma of the Gallbladder; Carcinoma of the Intrahepatic or Extrahepatic Biliary Tract; Xeloda; Eloxatin
MeSH Terms: conditions — Gallbladder Neoplasms; Biliary Tract Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + Oxaliplatin (Experimental): Combination of intravenous (IV) oxaliplatin 100 mg/m^2 Day 1 and oral (PO) capecitabine 750 mg/m^2 twice daily (total daily dose 1500 mg/m2) on Days 1-14.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — 1500 mg/m^2 PO twice daily x 14 days.
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m^2 IV over 2 hours on day 1 of cycle.
  Other Names: Eloxatin

SUMMARY:
This is a Phase II trial of the combination of oxaliplatin (Eloxatin) and capecitabine (Xeloda), known as XELOX, in participants with unresectable or recurrent cholangiocarcinoma, including carcinoma of the gallbladder or biliary tract, both intrahepatic and extrahepatic. Participants may be either previously untreated or treated with chemotherapy. Participants will accrue to two strata based on pre-treatment status; separate response rates and statistical operating characteristics will be applied to each stratum.

The primary objective is to determine the objective response rate (complete plus partial) of XELOX in this population.

Secondary objectives include determining toxicity, stable disease rates, and median and overall survival of participants treated with this combination.

DETAILED DESCRIPTION:
Oxaliplatin causes death of cancer cells and other actively dividing cells by interfering with DNA function. Capecitabine causes death of cancer cells by interfering with certain molecules that are important in cell division.

After the screening portion of the study, if you are eligible to continue, you will begin treatment with oxaliplatin and capecitabine. Once treatment begins, you will come to M. D. Anderson at least every three weeks (21 days) for treatment. Each 21-day period of treatment is called a "cycle" of therapy. You will receive at least 3 cycles of therapy unless side effects are severe or the cancer grows very quickly.

You will need to have a small tube (central venous line) inserted into a large vein under the skin of the chest or through a vein in the arm to receive oxaliplatin. The central venous line will remain in place the entire time you are taking part in this study. Oxaliplatin must be given at M. D. Anderson. On Day 1 of each cycle, you will receive oxaliplatin injected into a vein over 2 hours.

You will take capecitabine tablets by mouth 2 times a day for the first 2 weeks (Days 1-14) of each 3-week cycle. No treatment will be given for the last 7 days of each cycle (except if your first dose of capecitabine for a new cycle is taken in the evening, your last dose will be taken in the morning of Day 15.) You must take capecitabine within 30 minutes after breakfast and dinner. The morning and evening doses should be about 12 hours apart. You should take capecitabine with water, and not with fruit juices. At the first treatment visit and every 3 weeks, you will receive enough capecitabine to last until the next visit. At each visit, you must return any capecitabine you have not used as well as all empty bottles.

Before each new cycle of therapy, you will have a complete physical exam and blood (about 2 ½ teaspoons) will be collected for routine tests. You will be asked to tell the study doctor about all medications you have taken since you started taking the study drugs and any health problems that you may have experienced. During the first cycle, you will have a blood (about 2 teaspoons) sample collected each week for routine tests. You will also have either CT scans or a MRI of the tumor(s) every 9 weeks and at the end of the study. Additional tests may be done during the study if your doctor feels it is necessary for your care.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of the treatment. You may continue to receive treatment on this study until the disease gets worse or you experience any intolerable side effects. If this happens, you will be taken off the study and your doctor will discuss other treatment options with you.

When you stop taking part in the study, you will have blood (about 3 teaspoons) collected for routine tests. You will have a physical exam and either a CT scan or a MRI to check on the status of the disease. You will be contacted by phone every three months for the rest of your life to check on the status of the disease and on any symptoms you may be experiencing.

All tests before each new cycle of treatment and when treatment stops must be done at M. D. Anderson.

This is an investigational study. The drugs oxaliplatin and capecitabine are FDA approved for treatment of advanced cancer of the colon or rectum. However, the drugs are not approved for gallbladder or biliary tract cancer. Up to 50 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed carcinoma of the gallbladder, intrahepatic or extrahepatic biliary tract, not amenable to resection with curative intent.
* Participants must have measurable disease as per the modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria, defined as at least one lesion that can be accurately measured in at least one dimension, with minimum lesion size equal to or more than twice the slice thickness of the imaging study used.
* Participants who are previously untreated as well as those who have received prior therapy are eligible to participate in this study. Participants may have received up to a total of two prior chemotherapy regimens for their disease, including biologic therapy(ies). The same regimen may have been received at different times during the course of the Participant's treatment. Surgery, radiofrequency ablation, external beam radiotherapy, or other directed therapies do not count as prior regimens and are allowed.
* Previous treatment may include systemic chemotherapy, however, prior capecitabine (unless administered as a radiosensitizing agent concurrently with prior external beam radiotherapy) or oxaliplatin are excluded.
* If radiation was previously received, the measurable disease must be recurrent or metastatic disease outside the previous radiation field.
* A minimum of 4 weeks must have elapsed since completion of any prior chemotherapy or radiotherapy.
* Participants should have a life expectancy of at least 16 weeks based on the clinical judgment of the Investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 2 or Karnofsky > 70.
* Adequate bone marrow function defined as absolute peripheral granulocyte count of >/= 1500/mm3, platelet count >/= 100,000/ mm3, and hemoglobin >/= 10 gm/dL.
* Adequate renal function, defined as serum creatinine </= 1.5 times ULN institutional normal and calculated creatinine clearance >30 mL/min (using Cockcroft and Gault formula).
* Participants must have adequate hepatic function: total bilirubin </= 2.0 gm/dL; serum albumin >/= 2.5 gm/dL; transaminases up to 5 times the upper limit of institutional normal value; or prothrombin time prolonged up to 2 seconds greater than the institutional normal value.
* Negative serum pregnancy test in women with childbearing potential.
* The effects of the combination of oxaliplatin and capecitabine on the developing fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
* Participants must sign an Informed Consent and Authorization indicating that they are aware of the investigational nature of this study and the known risks involved.
* Age >/=18 years.
* Participants taking therapeutic dose-levels of coumarin-derivate anticoagulants should be switched to low Low molecular weight heparin (LMWH). Low-dose coumadin (e.g. 1 mg po per day) in Participants with in-dwelling venous access devices, is allowed.

Exclusion Criteria:

* Prior therapy with oxaliplatin or capecitabine; capecitabine administered as a radiosensitizing agent concurrently with prior external beam radiotherapy is allowable.
* Participants who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants may not be receiving any other investigational agents nor have received any investigational drug </= 30 days prior to enrollment.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical therapy affecting absorption.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Because Participants with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive Participants receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with XELOX. Appropriate studies will be undertaken in Participants receiving combination anti-retroviral therapy when indicated.
* Participants with extensive symptomatic fibrosis of the lungs.
* Peripheral neuropathy > grade 1.
* Known DPD deficiency.
* Participants receiving therapeutic doses of coumarin-derivative anticoagulant therapy are excluded since a drug interaction between capecitabine and coumarin anticoagulants has been reported. Participants requiring anticoagulation who may be safely switched to LMWH are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Thomas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: August 28, 2003 to July 31, 2006. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Following enrollment, one of the forty-four participants was found to be ineligible and never assigned to a group.
Groups:
- Capecitabine + Oxaliplatin: Combination of intravenous (IV) oxaliplatin 100 mg/m^2 Day 1 and oral capecitabine 750 mg/m^2 twice daily on Days 1-14.
Period: Overall Study
Arm/Group | Capecitabine + Oxaliplatin
Started | 44
Completed | 43
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 44
Age Continuous [Median (Full Range); unit: years] | 68 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective Response = Complete Response + Partial Response. Response evaluated using modification of new international criteria proposed by RECIST [changes in only largest diameter (unidimensional measurement) of tumor lesions used in the RECIST criteria]. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline with restaging every 3 cycles (cycle=21 days)
Population: Analysis was per protocol. One participant was found ineligible and received no treatment.
Measure: Number; unit: participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 43
participants | 1

ADVERSE EVENTS:
Time Frame: A total 3 years from August 2003 to December 2006.
Description: The subjects were provided a study calendar every cycle and instructed to record all side effects experienced.
Groups:
- Stratum: 1 Prior Regimen: Received prior therapy. Capecitabine + Oxaliplatin: Experimental. Combination of IV oxaliplatin 100 mg/m^2 Day 1 and oral capecitabine 750 mg/m^2 twice daily on Day 1-14.
- Stratum 2: No Prior Therapy: Previously untreated. Capecitabine + Oxaliplatin: Experimental. Combination of IV oxaliplatin 100 mg/m^2 Day 1 and oral capecitabine 750 mg/m^2 twice daily on Day 1-14.
Arm/Group | Stratum: 1 Prior Regimen | Stratum 2: No Prior Therapy
Serious Adverse Events (participants affected / at risk) | 4/18 | 2/26
Other Adverse Events (participants affected / at risk) | 18/18 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum: 1 Prior Regimen (N=18) | Stratum 2: No Prior Therapy (N=26)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) — Allergy/Immunology
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum: 1 Prior Regimen (N=18) | Stratum 2: No Prior Therapy (N=26)
Abdominal Pain (Gastrointestinal disorders) | 5 | 11
Alkaline Phosphatase (increase) (Hepatobiliary disorders) | 2 | 5
Anemia (Blood and lymphatic system disorders) | 2 | 4
Anorexia (Gastrointestinal disorders) | 4 | 14
Diarrhea (Gastrointestinal disorders) | 8 | 14
Dizziness (Nervous system disorders) | 0 | 6
Fatigue (General disorders) | 9 | 18
Flatulence (Gastrointestinal disorders) | 2 | 6
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 | 8
Headache (General disorders) | 4 | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 4
Jaw cramps (Musculoskeletal and connective tissue disorders) | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 9
Nausea (Gastrointestinal disorders) | 11 | 23
Neuropathy-sensory (Nervous system disorders) | 15 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Erythema multiform, Desquamation...) (Skin and subcutaneous tissue disorders) | 2 | 1
Serum Glutamic Oxaloacetic Transaminase (AST, SGOT) (Hepatobiliary disorders) | 3 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 4
Taste Disturbance (Gastrointestinal disorders) | 2 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 9
Vomiting (Gastrointestinal disorders) | 4 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No